CLINICAL TRIAL: NCT02665169
Title: Randomized Fall Prevention Trial For Aging Females by Providing Supervised Exercises and Free Use of Municipal Recreation Facilities.
Brief Title: Kuopio Fall Prevention Study.
Acronym: KFPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KUH5203083
Record Dates: First submitted 2016-01-11; First posted 2016-01-27 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Accidental Falls; Health Behavior; Aging
Keywords: Postural Balance; Cost-Benefit Analysis; Morbidity; Exercise
MeSH Terms: conditions — Health Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise intervention group (Experimental): Supervised exercise intervention of 12 months. One Taiji and one gym training per week for first six months followed by 6 months free independent use of municipal facilities, including gym, swimming hall and weight room. Written and oral health counselling provided.
  Interventions: Behavioral: Supervised physical exercise; Other: Health counselling
- Control group (Active Comparator): Control group, without any induced exercise intervention. Written and oral health counselling provided.
  Interventions: Other: Health counselling

INTERVENTIONS:
Behavioral: Supervised physical exercise — Supervised physical exercises in Taiji and weight training. Free use and access into municipal recreation and training facilities for one year.
  Arms: Exercise intervention group
Other: Health counselling — Health counselling, fall prevention strategies at home, information concerning municipal recreational services available.

SUMMARY:
This study evaluates the 6 month exercise intervention (Taiji and gym course) combined with free use of communal recreation facilities in fall prevention.

Morbidity, use of social services and health outcomes of aging women in province of Kuopio, Finland are also monitored. The study combines a six months supervised exercise, followed by six months free, but unsupervised, use of recreational facilities and observational period of second year into total of 2 year follow up duration.

DETAILED DESCRIPTION:
In 2016, a 2-year randomized controlled trial (RCT) will be launched to investigate the effect of exercise on fall risk, injuries and subjective well-being (SWB) in aging women (n=1078) by using municipal sport services in cooperation with the city of Kuopio. The effect of the exercise intervention on functional capacity, muscle strength, bone, body composition, cognitive function, the use of health services and its cost effectiveness will also be studied.

The trial will be carried out on women belonging to the Kuopio Osteoporosis Risk Factor and Prevention (OSTPRE) Study, which is an ongoing population-based prospective cohort study, with a follow-up of 26 years. It investigates life style factors associated with fractures falls, bone mineral density and morbidity in a target population of 14 220 women, now aged between 75-84 year.

The study combines combination of a 2-year fall prevention trial with the 26 years of life style and medical data from the previous OSTPRE follow up to provide meaningful answers whether municipal exercise program can provide cost effective health gain in elderly. In addition, the study aims to answer, who will benefit from the exercise the most and what are the underlying factors explaining efficacy in the women's previous 26 years of lifestyle and medical history. The study will help to develop strategies for societal fall prevention.

ELIGIBILITY:
Inclusion Criteria:

* Included in the previous Osteoprosis Risk Factors and Prevention (OSTPRE) study follow up protocol, conducted in Kuopio Finland, between 1989-2015.

Exclusion Criteria:

* Unstable angina pectoris, severe pulmonary disease, not self-ambulatory or institutionalized, moderate to severe dementia.

Ages: 75 Years to 84 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 914 (Actual)
Dates: Start 2016-03; Primary Completion 2019-05-30 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Risk of falls | Two years
  Method of assessment; Personal fall diary. In case of fall, subject records the event into logbook. Outcome: Number of Falls during follow up.
Risk of fall | Two years
  Biweekly text message (SMS) question concerning recent falls during last 2 weeks (Reply:Yes/No). In a case of a positive reply, following phone call to the subject to validate the event. Outcome: Number of Falls during follow up.

SECONDARY OUTCOMES:
Morbidity | two years
  Methods of assessment; Self reported health survey concerning chronic medical conditions. Outcome: Morbidity during follow up.
All cause morbidity | two years
  Methods of assessment; Use of national health care registries and hospital discharge registries. Outcome: Validated morbidity during follow up.
Functional capacity | two years
  Methods of assessment; Timed Get Up and Go Test (TUG). Outcomes; Time consumed the time that a person takes to rise from a chair, walk three metres, turn around, walk back to the chair, and sit down. Outcome: Time consumed in the task (Seconds).
Range of motion | two years
  Methods of assessment; Squatting test. Outcomes; Physical task to squat down, touch the floor with fingertips and get up, without additional support. Outcome: Able/unable to comply (Y/N).
Postural Balance | two years
  Methods of assessment; One leg stand test. Outcomes; Able to maintain static one leg standing position for ten second (Seconds), Outcome: able/unable to comply (Y/N).
Bone mineral density | two years
  Method of assessment; Dual X-ray Absorption (DXA) measurement in proximal femur. Outcomes; Areal bone mineral density (g/cm2).
Body composition | two years
  Method of assessment; Dual X-ray Absorption (DXA) total body scan. Outcomes; body soft tissue and bone mass distribution (g).
Grip strength | two years
  Methods of assessment; Maximal grip strength by using handheld dynamometer. Outcomes; Maximal muscle force produced (kg).
Leg muscle strength | two years
  Methods of assessment; isometric leg extension strength in a sitting position with a force plate device. Outcomes; Maximal muscle force produced (kg).
Muscle strength and balance | two years
  Methods of assessment; Balance test protocol by using force plate to measure body sway in various positions. Outcomes; velocity and distance of travel by the center of gravity (mm/second).
Depression | two years
  Methods of assessment; Geriatric Depression Scale (GDS). Outcomes: Units on a Scale
Life satisfaction | two years
  Methods of assessment; Life satisfaction scale (LS). Outcomes: Units on a Scale
Psychological stress | two years
  Methods of assessment; Perceived Stress Scale (PSS). Outcomes: Units on a Scale.
Psychological stress coping | two years
  Methods of assessment; Brief Resilience Coping Scale (BRCS). Outcomes: Units on a Scale.
Life orientation | two years
  Methods of assessment; Life Orientation Test (LOT-R) questionnaire Outcomes: Units on a Scale.
health-related quality of life (HRQoL) | two years
  Methods of assessment; 15-D self administered measure scale Outcomes: Units on a Scale.
Self perceived quality of life | two years
  Methods of assessment; World Health Organization WHOQOL-BREF. Outcomes: Units on a Scale.

OTHER OUTCOMES:
Life style habits | two years
  Self reported history of health behaviour by using OSTPRE study follow up data registry. Post hoc.
  Outcomes: Units on a scale.
Use of healthcare services | two years
  Use of health service use during the follow up by utilizing hospital discharge registries. Outcome: Resources spent in healthcare during follow up(Euros)

CONTACTS AND LOCATIONS:
Overall Officials: Heikki Kröger, Professor, Principal Investigator — Department of Surgery, Kuopio University Hospital; Toni Rikkonen, Dr, Principal Investigator — Kuopio Musculoskeletal Research Unit, University of Eastern Finland
Locations (1):
- Bone and Cartilage Research Unit, Clinical Research Centre, University of Kuopio, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tamminen AE, Honkanen R, Koivumaa-Honkanen H, Sirola J, Sund R, Kroger H, Rikkonen T. Exercise reduces the risk of falls in women with polypharmacy: secondary analysis of a randomized controlled trial. Sci Rep. 2025 Feb 19;15(1):6009. doi: 10.1038/s41598-025-88205-y. PMID 39972017
- [Derived] Vilpunaho T, Karinkanta S, Sievanen H, Kopra J, Kroger H, Rikkonen T. Predictive ability of a self-rated fall risk assessment tool in community-dwelling older women. Aging Clin Exp Res. 2023 Jun;35(6):1205-1212. doi: 10.1007/s40520-023-02423-w. Epub 2023 May 5. PMID 37145268
- [Derived] Vilpunaho T, Sund R, Koivumaa-Honkanen H, Honkanen R, Kroger H, Rikkonen T. Urban RCT participants were healthier than non-participants or rural women. J Clin Epidemiol. 2021 Dec;140:44-55. doi: 10.1016/j.jclinepi.2021.08.032. Epub 2021 Sep 3. PMID 34487834
- [Derived] Vilpunaho T, Kroger H, Honkanen R, Koivumaa-Honkanen H, Sirola J, Kuvaja-Kollner V, Sund R, Rikkonen T. Randomised controlled trial (RCT) study design for a large-scale municipal fall prevention exercise programme in community-living older women: study protocol for the Kuopio Fall Prevention Study (KFPS). BMJ Open. 2019 Jun 21;9(6):e028716. doi: 10.1136/bmjopen-2018-028716. PMID 31230026